CLINICAL TRIAL: NCT03764514
Title: Effectiveness of Spinal Cord Stimulation As Therapy for Chemotherapy-Induced Peripheral Neuropathy: a Pilot Trial
Brief Title: Spinal Cord Stimulation in Chemotherapy Induced Neuropathy
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00076097
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2023-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Spinal Cord Stimulator - Permanent Implantation
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — Permanent Implantation

SUMMARY:
This is an observational based pilot study evaluating the use of spinal cord stimulators for the treatment of chemotherapy induced peripheral neuropathy will lead to an increase in quality of life and decrease in pain.

DETAILED DESCRIPTION:
Cancer treatment, for many patients, results in painful side effects. As evidence mounts demonstrating the risks associated with long term opioid therapy, non-opioid modalities need to be developed. Spinal cord stimulators are implanted devices that modulate the pain signaling system in the spinal cord. This research hopes to determine if the use of a spinal cord stimulator in patients with chemotherapy induced peripheral neuropathy will lead to an increase in quality of life and decrease in pain.The primary endpoints will be the number of patients who undergo permanent implantation. The endpoints will measure pain with the Brief Pain Inventory Short Form visual analog scale. The sleep quality will be measured using the Pittsburgh Sleep Quality Assessment.

ELIGIBILITY:
Inclusion Criteria:

• The patient has persistent, severe peripheral neuropathy secondary to chemotherapy

Exclusion Criteria:

• Refusal to undergo a spinal cord stimulator procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Permanent Spinal Cord Stimulator Implantation | 2 years
  To determine the total number of patients who undergo permanent spinal cord stimulator implantation.

SECONDARY OUTCOMES:
Subjective Pain Assessment: Brief Pain Inventory-Short Form | 2 years
  Measure Pain with the Brief Pain Inventory-Short Form. The scale measures the severity of pain and the impact of pain on daily functions. The scale range includes 0-10 scales, with 0=no interference and 10=interferes completely. There is not a scoring algorithm, but "worst pain" or the average of the four severity items can be used as measures of pain severity; the average of the seven interference items can be used as a measure of pain interference.
Subjective Quality of Life Assessment: Pittsburgh Sleep Quality Assessment | 2 years
  Measure quality of life through the use of the Pittsburgh Sleep Quality Assessment. The Pittsburgh Sleep Quality Index is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations.The 19 items are grouped into 7 components, including (1) sleep duration, (2) sleep disturbance, (3) sleep latency, (4) daytime dysfunction due to sleepiness, (5) sleep efficiency, (6) overall sleep quality, and (7) sleep medication use. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (global score) indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Smith, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Patewood Memorial Hospital, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braun Filho JL, Braun LM. [Spinal cord stimulation in the treatment of refractory painful polineuropathy induced by chemotherapy.]. Rev Bras Anestesiol. 2007 Oct;57(5):533-8. doi: 10.1590/s0034-70942007000500008. Portuguese. PMID 19462129